CLINICAL TRIAL: NCT06378034
Title: Effect of Lactium on Sleep Efficiency and Quality in Healthy Volunteers With Persistent Subclinical Insomnia
Brief Title: Effect of Lactium on Sleep Disorders in Healthy Volunteers With Persistent Subclinical Insomnia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ingredia S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023-A01926-39
Record Dates: First submitted 2024-04-11; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactium (Active Comparator)
  Interventions: Dietary Supplement: Lactium
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactium — 300 mg per day, taken 30 min to 60 min before bedtime
  Arms: Lactium
Dietary Supplement: Placebo — 300 mg per day, taken 30 min to 60 min before bedtime
  Arms: Placebo

SUMMARY:
The main objective will be to assess the effect of Lactium® on sleep efficiency in volunteers presented with persistent subclinical insomnia.

ELIGIBILITY:
Inclusion Criteria:

* In good general and mental health according to the investigator judgement: no clinically significant and abnormalities relevant to medical history or clinical examination
* Having a Body Mass Index (BMI) of 18.5 < BMI < 30 kg/m2
* Present subclinical insomnia characterized by an Insomnia Severity Index (ISI) score between 8 and 14 during the last month preceding the screening visit
* Whose insomnia symptoms started at least 3 months before the screening visit
* Present a medium level of phycological stress characterized by a Perceived Stress Scale (PSS-10) score between 14 and 26
* Willing / able to maintain their eating habits and physical activity during the study (no planned diet, no change in physical activity ...)
* Willing / able to participate in the study in accordance with protocol procedures (dated and signed informed consent form)
* Affiliated to a Health insurance scheme
* Agree to be registered in the national database of subjects participating in clinical research
* Have a smartphone compatible with the NursTrial® e-PRO application

Exclusion Criteria:

1. Presenting moderate to severe insomnia defined by an ISI score greater than or equal to 15 in the last month prior to selection
2. Presenting other sleep disorders already diagnosed or suspected during the screening visit: impatience (restless legs), parasomnias, hypersomnias, sleep apnea, iatrogenic insomnia
3. Subject assessed as "definitely" an evening type people by the Horne and Ostberg's circadian typology questionnaire (delayed phase subject)
4. Whose sleep disorders are related to external factors (noise pollution, young children, etc ...)
5. Workers with atypical schedules (night work, staggered working hours, changes in regular working hours, or shift work)
6. Smoker
7. Drug Addict
8. Alcohol consumption greater than 2 glasses per day
9. Subject with excessive caffeine consumption exceeding 400 mg per day (coffee ≈ 80 mg per cup; cola soda≈ 25 mg per glass; tea ≈40 mg per cup; energy drinks ≈70 mg per glass)
10. Subject consuming or having consumed any dietary supplement with an effect or a possible effect on sleep, stress, anxiety, or fatigue during the last 3 months prior to screening visit (melatonin, lactium, ginseng, caffeine ...)
11. Subject who has been treated during the 6 months preceding the screening visit or are currently being treated with non-medication therapies (such as psychotherapy, Cognitive Behavioral Therapy [CBT], Eye Movement Desensitization and Reprocessing [EMDR], etc. or repetitive Transcranial Magnetic Stimulation [TMS]) or psychotropic medication prescribed and / or recommended for anxious manifestations, depression, sleep disorders and generally for any neurological or psychological manifestation
12. Subject with psychiatric comorbidity as described in the Diagnostic and Statistical Manual of Mental Disorders V (DSM-V) (depression, post traumatic stress disorder, etc.) or history of psychiatric illness
13. Untreated or not controlled hypertension
14. Untreated or not controlled thyroid diseases (hypo or hyperthyroidism, Graves' disease...)
15. Epileptic subject
16. Asthmatic subject
17. Any other pathology or medical history or symptomatology likely to significantly influence the study criteria (nocturnal pain, nasal congestion, cough at bedtime or nocturnal cough, nocturnal pollakiuria, tinnitus, etc.) according to the investigator
18. Confirmed cow's milk protein allergy
19. Sleeping on a mattress that is not compatible with the sleep quality recording (water and air mattresses) or does not have adequate or necessary domestic equipment for its operation (power socket near the bed, etc.)
20. Likely to sleep outside their home during the study (holidays, regular business trips, etc.)
21. Whose spouse or partner is participating in this study
22. Pregnant woman (negative urine test at screening and initial/randomization visits) or wishing to be pregnant during the study or breastfeeding
23. Hormonal state that may induce fluctuation in emotional state and sleep during the study, such as, the postpartum period (< 6 months after delivery) and perimenopause (irregular menstrual cycle, hot flashes)
24. Under legal protection (guardianship, curatorship) or deprived of rights following an administrative or judicial decision
25. Psychologically or linguistically incapable of understanding and signing informed consent
26. Participating in another clinical trial or in exclusion period of a previous clinical trial
27. Having reached the maximum research compensation threshold stipulated by regulations.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-10 (Estimated); Primary Completion 2024-07-15 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Sleep efficiency | Before treatment (day 0); at the end of the treatment (after 29 days)
  The primary endpoint will be changes between baseline and final sleep efficiency (SE), measured nightly using actigraphy

SECONDARY OUTCOMES:
Sleep diary | Before treatment (day 0); at the end of the treatment (after 29 days)
  Changes between baseline and final subjective sleep quality parameters, recorded in the sleep diary
Insomnia Severity Index | Before treatment (day 0); at the end of the treatment (after 29 days)
  Changes between the baseline and intermediate and final values of the Insomnia Severity Index (ISI) total score Present subclinical insomnia characterized by an Insomnia Severity Index (ISI) score between 8 and 14 e. The sub-scores of the ISI correspond to 0-7: Lack of insomnia, 8-14: Subthreshold (=subclinical) insomnia, 15- 21: Moderate insomnia, 22-28: Severe insomnia.
PSQI | Before treatment (day 0); at the end of the treatment (after 29 days)
  Changes between the baseline and final values of Pittsburgh Sleep Quality Index (PSQI) total score Score 0: no sleep diroders, >5 moderate sleep disorders; 21: severe sleep disorders
Sleep quality by cctigraphy | Before treatment (day 0); at the end of the treatment (after 29 days)
  Changes between baseline and final objective sleep quality by actigraphy